CLINICAL TRIAL: NCT07162207
Title: Evaluation of Pinhole Technique Using Bi-layer Collagen Membrane Versus Subepithelial Connective Tissue Graft in the Treatment of Localized Gingival Recession: A Randomized Clinical Trial
Brief Title: Bi-layer Collagen Membrane Versus Subepithelial Connective Tissue Graft in the Treatment of Localized Gingival Recession
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Aya Elleithy, Assistant lecturer of Oral Medicine and Periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-REC 052317
Record Dates: First submitted 2025-08-21; First posted 2025-09-09 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Gingival Recession, Localized
Keywords: Gingival recession; pinhole surgical technique; Connective tissue graft; Bi-layer collagen membrane
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sub Epithelial Connective tissue graft (Active Comparator): A pinhole is created in the site of recession. After harvesting the connective tissue graft from the palate it's trimmed and inserted in the tunnel.
  Interventions: Procedure: Pinhole surgical technique
- Bi-layer collagen membrane (Experimental): A pinhole is created in the site of recession, the Bi-layer collagen membrane is trimmed to fit the size of the recession defect, followed by membrane insertion in the tunnel.
  Interventions: Procedure: Pinhole surgical technique

INTERVENTIONS:
Procedure: Pinhole surgical technique — A pinhole is created in the site of recession, the grafting material (Bi-layer collagen membrane versus connective tissue graft) is trimmed to fit the size of the recession defect, followed by graft insertion in the tunnel.

SUMMARY:
The goal of this clinical trial is evaluation of the change in depth and width of gingival recession in terms of gingival thickness and esthetics, and evaluation of patient satisfaction in terms of postoperative pain and final esthetic appearance.

The study will be conducted on twelve Egyptian healthy patients with localized gingival recession. Researchers will compare clinical effectiveness of collagen membrane to connective tissue graft in treatment of localized gingival recession. The study hypothesis is that no difference exists between Bilayer collagen membrane combined with Pinhole approach and CT graft combined with Pinhole approach used for root coverage in treatment of localized gingival recession.

DETAILED DESCRIPTION:
Twelve patients with localized gingival recession were randomly assigned into two equal groups. The control group received treatment with Pinhole surgical approach using connective tissue graft material, while the comparison group received treatment with Pinhole surgical approach using collagen membrane. Patients were followed up after 3 and 6 months from treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have ages above 18 years.
2. Patients included in the study are classified with Cairo RT1 and RT2 localized recession defect Cairo et al. (2011).
3. Patients have at least 1 mm of residual keratinized tissue.
4. Recession depth ≥ 2mm.
5. Recession is not caused by periodontal disease.
6. Patients have good oral hygiene.

Exclusion Criteria:

1. Patients with systemic diseases.
2. Pregnant and lactating women.
3. Smoking patients and drug abusers.
4. Patients with mal-positioned and rotated teeth.
5. Patients with periodontally affected teeth adjacent to the treated sites.
6. Patients having carious lesions or restorations in the treated teeth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
The change in depth of gingival recession (RD) | The change from enrollment to 24 weeks.
  -This clinical parameter will be measured to evaluate the primary outcome: (unit of measurement: millimeters).
  - This parameter will be recorded at baseline (just prior to the surgery) as well as at the 3rd month and 6th month follow up for Group 1 and Group 2.
The change in the width of gingival recession. | The change from enrollment to 24 weeks.
  This clinical parameter will be measured to evaluate the primary outcome: (unit of measurement: millimeters).
  - This parameter will be recorded at baseline (just prior to the surgery) as well s at the 3rd month and 6th month follow up for Group 1 and Group 2.
Plaque index (PI): | This parameter is measured at baseline, 3 and 6 months postoperatively.
  - Plaque index is based on recording both soft debris and mineralized deposits for each surface of the teeth (buccal, lingual, mesial and distal). Each of the four surfaces of the teeth is given a score from 0-3.
Gingival index (GI) | This parameter is measured at baseline, 3 and 6 months postoperatively.
  - Gingival index is measured by giving a score from 0-3 for each surface of the four surfaces of the tooth then divided by four to give gingival index of each tooth.
Probing depth (PD) | This parameter will be recorded at baseline, 3 and 6 months postoperatively.
  - Probing depth is measured from the gingival margin to the depth of the gingival sulcus using UNC-15 periodontal probe at 6 sites for each tooth: mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual and disto-lingual surface.
Clinical attachment level (CAL) | CAL will be measured at baseline, 3 and 6 months postoperatively.
  - Clinical attachment level is measured from the cemento-enamel junction (CEJ) to the depth of the gingival sulcus.
Percentage of mean root coverage (MRC %) | MRC% is recorded at baseline, 3 and 6 months postoperatively.
  Percentage of mean root coverage is calculated as: ([RD preoperative - RD postoperative]/ RD preoperative) × 100 % (unit of measurement: Percentage % ).
Width of keratinized tissue (KTW) | This parameter is measured at baseline, 3 and 6 months postoperatively.
  Width of keratinized tissue (KTW) is measured from the most apical extension of gingival margin to the mucogingival line.
Gingival thickness (GT) | This parameter is recorded at baseline, 3 and 6 months postoperative.
  Gingival thickness (GT) is measured using UNC-15 periodontal probe with piercing the mucosal surface at a right angle with slight pressure until reaching the hard tissue. The distance between the tip of the probe and the outer mark is measured.

SECONDARY OUTCOMES:
Evaluation of patient satisfaction in terms of post-operative pain. | assessment at one week postoperative time.
  It's assessed by using verbal, numeric scale and by recording amount of analgesic intake postoperatively. The Visual Analogue Scale (VAS) pain score: is a psychometric response to pain reported by the patient directly through a score (between 0 and 10. 0: no pain, 1: minimal pain, 5: moderate pain, 10: severe pain). This was done through a questionnaire 1st week after surgery. Post-operative pain was assessed indirectly by mean consumption of analgesics for 7 days postoperatively.
Evaluation of patient satisfaction in terms of final esthetic appearance. | The change from enrollment to 24 weeks
  The clinical parameter: Root coverage esthetic score (RES) will be measured to evaluate the secondary outcome, time of evaluation at 6 months follow up time.
  - It is used to evaluate five variables and recorded at 6 months following surgery; these variables are gingival margin (GM), marginal tissue contour (MTC), soft tissue texture (STT), MCJ alignment and gingival color (GC). Then; giving score for each variable and added them to give score as the following GM: zero points= failure of root coverage (gingival margin apical or equal to the baseline recession); 3 points= partial root coverage; 5 points= Complete root coverage (CRC). MTC, STT, MGJ, GC are given zero point and 1 point according to certain criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Hala A. Abu El-Ela, Professor, Study Director — Faculty of Dentistry- Ain Shams University
Locations (1):
- Faculty of Dentistry- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pubmed in a database that has been used globally for research purposes — https://pubmed.ncbi.nlm.nih.gov/